CLINICAL TRIAL: NCT01072552
Title: Effect of Palivizumab Treatment on Subsequent Recurrent Wheezing in Preterm Infants: Case-control Study by Scientific Committee of Recurrent Wheezing (SCREW)
Brief Title: Effect of Palivizumab on Later Recurrent Wheezing in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Satoshi Kusuda (Other)
Collaborators: Scientific Committee of Recurrent Wheezing (Network)
Responsible Party: Sponsor-Investigator, Satoshi Kusuda, Professor of Neonatology, Tokyo Women's Medical University
Organization: Tokyo Women's Medical University (Other)
Other Study IDs: SCREW-001
Record Dates: First submitted 2009-12-21; First posted 2010-02-22 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Wheezing; Wheezing; Asthma
Keywords: recurrent wheezing; asthma; preterm infants; palivizumab; atopic diseases
MeSH Terms: conditions — Respiratory Sounds; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treated: Palivizumab treated
- Untreated: Palivizumab untreated

SUMMARY:
The hypothesis of the present study is that the prophylaxis with palivizumab to prevent the severe RS virus infection during the infancy among preterm infants may reduce the risk of subsequent recurrent wheezing in childhood.

The infants born between July 1st and December 31st in 2007 with the gestational age between 33 and 35 weeks were enrolled into the study at the end of RS virus infection season, April 2008. The infants were unintentionally divided into two groups, either palivizumab treated or untreated group at the enrollment, because the timing for palivizumab prophylaxis were already ended.

The study infants will be followed up until the age of 3 with recording the incidence of either parent reported or physician diagnosed recurrent wheezing.

The difference of the incidence of the recurrent wheezing between the groups will be analyzed with Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Infants born July ~ December 2007 at 33~35 weeks of gestation

Exclusion Criteria:

* Intrauterine growth retardation (less than -2.5SD)
* Infants with chronic lung disease (CLD) or other respiratory disease
* Infants received mechanical ventilation.
* Infants with chronic heart disease (CHD) or congenital anomaly (such as immunodeficiency).
* Infants received less than 3 doses of palivizumab during the first 6 months of life

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with the gestational age between 33 and 35 weeks
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of recurrent wheezing confirmed by physicians | two years

SECONDARY OUTCOMES:
Cumulative incidence of recurrent wheezing confirmed by parents | two years
Incidence of atopic asthma evaluated by SCREW according to the results of the questionnaire and hematological examination | two years
Cumulative incidence of wheezing confirmed by parents | two years
Cumulative incidence of wheezing confirmed by physicians | two years
Number of hospital/clinic visits and hospitalizations due to respiratory-related diseases | two years

CONTACTS AND LOCATIONS:
Overall Officials: Sankei Nishima, MD, Study Director — National Fukuoka Hospital; Kenji Okada, MD, Principal Investigator — National Fukuoka Hospital
Locations (1):
- Tokyo Women's Medical University, Shinjuku, Tokyo, Japan

REFERENCES:
- [Derived] Yoshihara S, Kusuda S, Mochizuki H, Okada K, Nishima S, Simoes EA; C-CREW Investigators. Effect of palivizumab prophylaxis on subsequent recurrent wheezing in preterm infants. Pediatrics. 2013 Nov;132(5):811-8. doi: 10.1542/peds.2013-0982. Epub 2013 Oct 14. PMID 24127479